CLINICAL TRIAL: NCT00863317
Title: A Randomized, Double Blind, Placebo Controlled Trial of Daily Montelukast for the Treatment of Viral Bronchiolitis
Brief Title: Trial of Montelukast for Treatment of Acute Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Frank Petruzella, Pediatric Emergency Physician, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDP-01; IND 103263 (Other: FDA)
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; montelukast; leukotriene inhibitor
MeSH Terms: conditions — Bronchiolitis | interventions — montelukast; Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- montelukast sodium (Experimental): 4mg granules PO QD for 14 days
  Interventions: Drug: montelukast sodium
- Placebo (Placebo Comparator): Sucrose granules PO QD for 14 days
  Interventions: Other: sucrose

INTERVENTIONS:
Drug: montelukast sodium — 4mg granules daily for 14 days
  Other Names: singulair
  Arms: montelukast sodium
Other: sucrose — table sugar as placebo daily for 14 days
  Arms: Placebo

SUMMARY:
The primary rationale for this study is to evaluate the effect of once daily montelukast on duration of acute illness in infants with first-time bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants aged 3 to 12 months of age
* Diagnosis by emergency physician of bronchiolitis

Exclusion Criteria:

* Any previous episode, as determined by a physician, of wheezing, bronchiolitis or asthma
* Any history of previous bronchodilator use prior to this illness
* Treatment with corticosteroids in the 14 days prior to the current illness
* Immunosuppression
* Immunodeficiency
* Caregiver does not speak English
* Diagnosis by the treating ED physician of croup
* Diagnosis by the treating ED physician of pneumonia
* Caregiver does not have access to a telephone

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gorelick, MD, MSCE, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast: 4mg granules
  montelukast sodium: 4mg granules daily for 14 days
Period: Overall Study
Arm/Group | Montelukast | Placebo
Started | 68 | 73
Completed | 60 | 64
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Sucrose | Total
Number analyzed (Participants) | 60 | 64 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 64 | 124
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 32 | 35 | 67
Region of Enrollment [Number; unit: participants]
  United States | 60 | 64 | 124

OUTCOME MEASURES:

1. Primary Outcome: Duration of Cough
Time Frame: up to 4 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 60 | 64
days | 13 [1 to 45] | 11 [2 to 63]

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Assessment was made via weekly follow up telephone interviews
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/73
Other Adverse Events (participants affected / at risk) | 7/68 | 5/73
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=68) | Placebo (N=73)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes